CLINICAL TRIAL: NCT05379439
Title: Family Connections: Structured Family Deliberation for Decisions About Home Ventilation
Brief Title: Family Connections
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB protocol was terminated
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00323418
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Chronic Respiratory Failure
Keywords: Tracheostomy; Home mechanical ventilation; Children with medical complexity; Medical ethics; Qualitative research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention families will participate in the Structured Family Deliberation that includes a clinician-led review of a web-based decisional aid.
  Interventions: Other: Structured Family Deliberation
- Control (No Intervention): Control families will undergo the standard decisional process for home ventilation and will also review the web-based decisional aid independently.

INTERVENTIONS:
Other: Structured Family Deliberation — Intervention families will be guided through the six modules included in the web-based decisional aid using a Structured Family Deliberation Tool. Parents will view narrated videos corresponding to each module and will be asked a series of questions related to their own lives and values. The process will continue until all modules are reviewed and all questions are completed.
  Arms: Intervention

SUMMARY:
This study seeks to evaluate a Structured Family Deliberation that will serve as the primary intervention in a multicenter controlled trial involving families considering tracheostomy and home ventilation for the child. In this study, the investigators will evaluate the feasibility, usefulness, face validity, and preliminary impact of this approach on preparedness for decision making among participants.

DETAILED DESCRIPTION:
The investigators will recruit 10 intervention families and 5 control families who are currently admitted to the neonatal or pediatric intensive unit and whose physician anticipates a decision about home ventilation within the next 30 days. Intervention families will receive the Structured Family Deliberation, which includes a guided review of a web-based decisional aid. Control families will receive a link to the website for independent review. All families will be assessed at 1 month with a survey assessing preparedness for decision-making, parental stress and coping, and a qualitative interview.

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians of children admitted to the neonatal or pediatric intensive care unit and whose physician anticipates a decision about home ventilation within the next month.

Exclusion Criteria:

* Parents will be excluded if:
* their child is in foster care or state guardianship
* they are unable to understand the purpose of the study
* they cannot reasonably participate in study demands
* are not fluent in English (the web-based decisional aid is not yet available in other languages).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by proportion of families enrolled | Duration of study period (12 months)
  Feasibility will be measured by the proportion of families approached that are successfully enrolled.
Feasibility as assessed by time spent engaging with the website by parents | Assessed at 30 day follow-up interview
  Feasibility will be measured by time parents spend engaging with the website.
Feasibility as assessed by proportion of successfully completed interventions | Duration of study period (12 months)
  Feasibility will be measured by success completing the intervention by the study team

SECONDARY OUTCOMES:
Usefulness of the Structured Family Deliberation Process will be assessed by participant responses to qualitative interview questions | Assessed at 30 day follow-up interview
  Qualitative interviews will be used to determine whether participants perceived either process as useful.
Preparedness in decision making as assessed by Preparation for Decision-Making Scale | Assessed at 30 day follow-up interview
  Preparation for decision-making will be assessed using a validated survey (Preparation for Decision-Making Scale). Scores range from 10-50; A higher score on the Preparation for Decision-Making scale indicates greater preparedness.
Factors in decision making as assessed by participants responses to qualitative interview questions | Assessed at 30 day follow-up interview
  Preparation for decision-making will be assessed by a qualitative interview with each family.
Parental stress and coping as assessed by participants responses to qualitative interview | Assessed at 30 day follow-up interview
  Parental stress and coping will be assessed assessed by a qualitative interview with each family.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Jabre, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States